CLINICAL TRIAL: NCT02640378
Title: Semiquantitative Urine Pregnancy Test Results At ≥9 Weeks of Gestation
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 1018
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: NO intervention — This study was a cross-sectional study. It had no intervention.

SUMMARY:
Purpose of study is to obtain data on urinary HCG concentrations at >9 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* pregnant at >9 weeks of gestation

Exclusion Criteria:

* none

Ages: 10 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: pregnant women at >9 weeks gestation
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2014-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Urine HCG concentration | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Raymond, Study Director — Gynuity Health Projects

IPD SHARING:
Plan to Share IPD: No